CLINICAL TRIAL: NCT07332650
Title: Prospective Clinical Investigation to Evaluate the Safety and Performance of Poly-L-lactic Acid - Juläine™ in Improving Gluteal Skin Laxity in Adults
Brief Title: Prospective Clinical Investigation to Evaluate the Safety and Performance of Juläine™ in Improving Gluteal Skin Laxity in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordberg Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NB 15-TF-BZ-100-08F
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Skin Quality; Skin Laxity
Keywords: Poly-L-lactic acid; PLLA; Aesthetic; Injectable filler; Buttocks; Gluteal skin laxity; Buttock skin laxity; Skin elasticity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate-treatment group (Experimental)
  Interventions: Device: Poly-L-Lactic Acid (Juläine™)
- Delayed-treatment group (delayed-start control) (Other)
  Interventions: Device: Poly-L-Lactic Acid (Juläine™)

INTERVENTIONS:
Device: Poly-L-Lactic Acid (Juläine™) — Juläine™ is a sterile injectable medical device composed of polylactic acid microspheres.

SUMMARY:
This study aims to evaluate the efficacy and safety of Juläine™ (poly-L-lactic acid) intradermal injections for the treatment of mild to moderate buttock skin laxity. Participants will be randomized to an immediate-treatment group or a delayed-treatment group. The immediate-treatment group will receive 2 to 3 treatment sessions over up to 2 months and will be compared with the delayed-treatment group during the control period; the delayed-treatment group will receive the same treatment after the delay. The primary objective is to assess clinical improvement in buttock skin elasticity 6 months after the last treatment, defined as an increase in global skin elasticity measured by a cutometer. Total study participation is up to 16 months, including follow-up. This multicenter trial will be conducted in Brazil.

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomized, parallel-group clinical investigation conducted in Brazil to evaluate the efficacy and safety of Juläine™ (poly-L-lactic acid) administered as intradermal injections for the treatment of mild to moderate skin laxity in the buttock (gluteal) region in adults.

A total of 90 participants will be randomized to either an immediate-treatment group or a delayed-treatment group (delayed-start control). Participants in the immediate-treatment group will receive Juläine™ intradermal injections in up to three sessions at Day 0, Day 30, and Day 60. During this initial control period, outcomes in the immediate-treatment group will be compared with those in the delayed-treatment group, which will not receive treatment. After the control period, participants in the delayed-treatment group will receive the same Juläine™ regimen at Day 240, Day 270, and Day 300. Each participant will remain in the study for up to 16 months, including screening, treatment sessions, and follow-up assessments.

The primary efficacy endpoint is improvement in buttock skin elasticity 6 months after the last treatment, defined as an increase in global skin elasticity measured by a cutometer, with assessments at screening/baseline and at the primary post-treatment timepoint. The mean change in global skin elasticity measured by cutometer, Global Aesthetic Improvement Scale (GAIS), and BODY-Q will also be evaluated, comparing groups during the control period.

Safety will be monitored through the collection of adverse events (AEs) through 240 days after treatment initiation, with comparisons between groups during the control period. Adverse events will also be evaluated through extended follow-up, including up to 180 days in the overall study population and up to 480 days in the immediate-treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 55 years;
* Body Mass Index (BMI) up to 25 kg/m²;
* Mild to moderate skin laxity in the gluteal region;
* Ability to understand the study and provide informed consent, attend follow-up visits, and follow post-injection instructions.

Exclusion Criteria:

* Pregnancy or breastfeeding, or planned pregnancy/lack of adequate contraception (through 8 weeks post-study);
* Active infection/inflammation near the treatment site or acute infection at screening;
* Severe/very severe gluteal skin laxity;
* Autoimmune disease or immunodeficiency;
* History of hypertrophic scarring/keloids or impaired wound healing risk;
* Prior buttock surgery or buttock aesthetic procedures within 6 months; planned/ongoing buttock-area aesthetic procedures during the study.
* Bleeding disorder/ongoing anticoagulant therapy;
* Recent systemic corticosteroids/immunosuppressants (past 2 months) or other collagen-inhibiting agents;
* Known hypersensitivity to investigational product components;
* Significant dermatologic/systemic disease (e.g., recurrent herpes simplex, skin malignancy);
* Planned weight-loss treatment during the study;
* Any other medical or psychological condition that, in the investigator's opinion, could interfere with study participation or with the assessment of outcomes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve an improvement in gluteal skin elasticity | Baseline and 180 days after completion of treatment.
  Proportion of participants who achieve an improvement in gluteal skin elasticity 6 months after the last treatment with Juläine™, predefined as an increase in global skin elasticity measured by cutometer.

SECONDARY OUTCOMES:
Mean change in global medial skin elasticity | Baseline and 180 days after completion of treatment.
  Mean change in global medial skin elasticity measured by cutometer 180 days after treatment completion.
Global improvement based on Global Aesthetic Improvement Scale (GAIS) evaluated by investigator and patient | Baseline and 180 days after completion of treatment.
  Proportion of participants with improvement on investigator and patient-rated Global Aesthetic Improvement Scale (GAIS) 180 days after treatment completion.
  The GAIS scale values are:
  1. Very much improved
  2. Much improved
  3. Improved
  4. No change
  5. Worse
  Where 1 represents the best outcome and 5 represents the worst.
Proportion of participants with improvement in BODY-Q score | Baseline and 180 days after completion of treatment
  Proportion of participants with improvement in BODY-Q score 180 days after treatment completion.
  The BODY-Q Buttocks scale is a patient-reported outcome (PRO) instrument designed to assess:
  -Satisfaction with the body appearance and quality of life.
  Each item is rated using a Likert-type response scale. Example response options include:
  * Very dissatisfied;
  * Dissatisfied;
  * Satisfied;
  * Very satisfied.
  Each response is assigned a numeric value. The raw score is then transformed using the BODY-Q scoring algorithm (Rasch-based) into a 0-100 scale.
  Where higher values reflect greater satisfaction.